CLINICAL TRIAL: NCT02420509
Title: Phase II Study to Evaluate Postoperative Chemotherapy in High-Grade Appendiceal Adenocarcinoma With Peritoneal Carcinomatosis
Brief Title: Postoperative Chemotherapy in High-Grade Appendiceal Adenocarcinoma With Peritoneal Carcinomatosis
Status: Terminated | Type: Observational
Why Stopped: unable to accrue
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joel Baumgartner, Assistant Professor of Surgery, University of California, San Diego
Other Study IDs: 150295
Record Dates: First submitted 2015-04-14; First posted 2015-04-20 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Neoadjuvant Therapy; Fluorouracil; Leucovorin; Capecitabine; Bevacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- systemic chemotherapy after CRS/HIPEC: Single-arm, prospective study of systemic chemotherapy after CRS/HIPEC. Subjects will be given twelve months of 5-FU or capecitabine with bevacizumab starting 4-8 weeks after surgery. CTRI Biostatistics Core personnel will assist in conducting analyses using the latest version of R (R Foundation for Statistical Computing, Vienna, Austria. http://www.R-project.org/).
  Interventions: Drug: systemic chemotherapy

INTERVENTIONS:
Drug: systemic chemotherapy — twelve months of 5-FU or capecitabine with bevacizumab starting 4-8 weeks after surgery
  Other Names: 5-FU; LEUCOVORIN; CAPECITABINE; BEVACIZUMAB

SUMMARY:
The purpose of this study is to find out if postoperative chemotherapy in patients with high-grade appendix cancer after surgery improves outcomes.

The postoperative chemotherapy will consist of 5-FU (with leucovorin) or capecitabine with bevacizumab. These drugs are approved for use in people with colon cancer, and they are used at UCSD for some patients with appendix cancer.

The purpose of this study is to explore the safety and efficacy of the postoperative chemotherapy treatment on cancer.

DETAILED DESCRIPTION:
This is an observational, single-cohort, prospective study of systemic chemotherapy after CRS/HIPEC. Subjects will be given twelve months of 5-FU or capecitabine with bevacizumab starting 4-16 weeks after surgery. CTRI Biostatistics Core personnel will assist in conducting analyses using the latest version of R (R Foundation for Statistical Computing, Vienna, Austria. http://www.R-project.org/).

No therapy is included in this study. Subjects have already previously undergone surgery for their cancer. This study will observe the outcomes of the postoperative chemotherapy treatment the doctor chooses to treat the subject's cancer.

ELIGIBILITY:
3.1 Inclusion Criteria Patients must meet all of the inclusion criteria to participate in this study.

1. Ability to understand and the willingness to sign a written informed consent.
2. High-grade peritoneal carcinomatosis from appendiceal adenocarcinoma.

   1. Moderate or poorly-differentiated adenocarcinoma, signet ring cell carcinoma or "high-grade" carcinoma (in primary tumor or extra-appendiceal metastases) as designated by standardized pathologic testing.23,24
   2. May be initially determined from pre-CRS/HIPEC tumor pathology (for screening purposes), but must be confirmed with pathology from resected tumors as part of CRS/HIPEC.
3. Have had complete (CC-0 or CC-1) CRS with HIPEC open or minimally invasive (laparoscopic or robotic)
4. Have received or plan to receive 12 months of postoperative chemotherapy, starting no sooner than 4 weeks and no longer than 16 weeks after CRS/HIPEC, consisting of:

   1. 5-fluorouracil (Adrucil®) 400 mg/m2 IV bolus then 2400 mg/m2 IV continuous infusion x 46hrs, leucovorin (Leucovorin Calcium) 20 mg/m2 IV bolus and bevacizumab (Avastin®) 5 mg/kg IV every two weeks for a total of 12 months (26 cycles); OR
   2. Capecitabine (Xeloda®) 1250 mg/m2 PO twice daily for 14 days, with 7-day break, bevacizumab (Avastin®) 7.5 mg/kg IV every three weeks, for a total of 12 months (17 cycles).
5. Have received or plan to receive standard clinical, biochemical and radiographic surveillance, consisting of:

   1. Adverse event assessments every chemotherapy cycle and at the end of treatment
   2. CEA, CA19-9 and CA 125

   i) Every 1 month x 1 year (during treatment), then ii) Every 1 month x 6 months, then iii) Every 3 months x 1.5 years, then iv) Every 6 months x 1 year c) CT chest, abdomen and pelvis or MRI i) Every 3 months x 1 year (during treatment), then ii) Every 3 months x 1 year, then iii) Every 6 months x 1 year, then iv) Every 12 months x 1 year
6. Age > 18 years old
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 (Appendix A).
8. Adequate organ and bone marrow function as defined below:

   1. Absolute Neutrophil Count ≥ 1.5 x 109/L
   2. Platelet count ≥ 100 x 109/L
   3. Hemoglobin ≥ 9.0 g/dL
   4. Total bilirubin ≤ 1.5 x ULN
   5. AST/SGOT and ALT/SPGT ≤ 2.5 X ULN
   6. Serum creatinine ≤ 1.5 x ULN
9. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

   a) A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: i) Has not undergone a hysterectomy or bilateral oophorectomy; or ii) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
10. Women of child-bearing potential must have negative pregnancy test prior to initiating study drug treatment.

3.2 Exclusion Criteria Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

1. Current or anticipated use of other investigational agents.
2. Patients who have received systemic chemotherapy or radiotherapy within two months prior to first scheduled cycle of postoperative chemotherapy.
3. Patients who are less than 4 weeks from CRS/HIPEC or have insufficient recovery from surgical-related trauma or wound healing as determined by the patient's surgeon.
4. History of hypersensitivity reaction specifically attributed to compounds of similar chemical or biologic composition to 5-FU, leucovorin, capecitabine or bevacizumab.
5. History of deep venous thrombosis (DVT) or pulmonary embolism (PE).
6. Concurrent active or measurable malignancies, except basal cell carcinoma or squamous cell carcinoma of the skin.
7. Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
8. Known diagnosis of human immunodeficiency virus (HIV) infection.
9. Incarcerated patients.
10. Pregnant or nursing women, due to the potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are those with peritoneal carcinomatosis secondary to high-grade appendiceal cancer who have undergone complete cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC), open or minimally invasive (laparoscopic or robotic), who plan to receive 12 months of 5-fluorouracil OR Capecitabine (Xeloda®), with Bevacizumab (Avastin®) for 12 months, with biochemical and radiologic surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 4 years
  PFS will be measured from the time of the start of postoperative chemotherapy until disease progression or death during the total study period (four years)

SECONDARY OUTCOMES:
Overall Survival | 4 years
  OS will be measured from the time of the start of postoperative chemotherapy until death during the total study period (four years)
Safety and Feasibility | Safety and feasibility of the chemotherapy regimen will be measured from the time of the start of postoperative chemotherapy until completion of chemotherapy (one year)
  Safety and feasibility of the chemotherapy regimen will be measured from the time of the start of postoperative chemotherapy until completion of chemotherapy (one year)
Quality of life will be measured by the Functional Assessment of Cancer Therapy | Quality of life will be measured from prior to surgery until study completion (four years)
  Quality of life will be measured by the Functional Assessment of Cancer Therapy, Colorectal Symptom Index (FCSI).

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Baumgartner, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No